CLINICAL TRIAL: NCT04466865
Title: Best Case/Worst Case: A Multisite Randomized Clinical Trial of Scenario Planning for Patients With End-Stage Kidney Disease
Brief Title: A Communication Tool to Assist Older Adults Facing Dialysis Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Pittsburgh (Other); University of Vermont (Other); Johns Hopkins University (Other); University of Colorado, Denver (Other); Icahn School of Medicine at Mount Sinai (Other); University of Washington (Other); West Virginia University (Other); Columbia University (Other); Medical College of Wisconsin (Other); The Palliative Care Research Cooperative Group (Unknown); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022-0193; 1R01AG065365-01 (NIH); A539750 (Other: UW, Madison); SMPH/SURGERY (Other: UW, Madison); Protocol Version 1/23/2025 (Other: UW Madison); 2019-1074 (Other: UW Madison)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Palliative Care; Kidney Failure, Chronic; Decision Making; Decision Support Techniques; Renal Dialysis; Dialysis; Kidney Diseases; Nephrologists; Decision Aid; End of Life; End-Stage Renal Disease; Late-Stage Renal Disease; Communication; Life-Supporting Treatments
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Death; Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Case/Worst Case communication tool (Experimental): The participant's enrolled nephrologist will have completed training on the Best Case/Worst Case communication tool and will be encouraged to use it with the participant.
  Interventions: Other: Best Case/Worst Case communication tool training
- Usual Care (No Intervention): Usual care conversations are typically focused on mode and timing of dialysis, management of electrolytes and scheduling of laboratory testing. Conservative management or a treatment option of "no dialysis" is rarely mentioned.

INTERVENTIONS:
Other: Best Case/Worst Case communication tool training — The communication tool promotes dialogue and patient deliberation, and supports shared decision making in the context of kidney disease. Building on a conceptual model of shared decision-making proposed and the practice of scenario planning the intervention is designed to lead to a discussion of participants preferences and consideration of outcomes.
  The nephrologist verbally describes the "best case," "worst case," and "most likely" outcomes for each treatment option-incorporating rich narrative from clinical experience and translation of probabilistic information-while drawing a diagram of those options. The nephrologist also writes details about each option on the diagram. The narrative and graphic help family and patients formulate and express preferences.
  Arms: Best Case/Worst Case communication tool

SUMMARY:
The purpose of this study is to test the effect of the "Best Case/Worse Case" (BC/WC) communication tool on receipt of palliative care and intensity of treatment at the end of life, quality of life, and quality of communication for older patients with end-stage renal disease (ESRD) receiving outpatient care at ten nephrology clinics. The intervention was developed and tested with acute care surgical patients at the University of Wisconsin (UW) and is now being testing to see if the intervention will work in a different setting.

The intervention will be tested with 320 older adults who have end-stage renal disease (ESRD) and are receiving care from a nephrologist enrolled in the study. Randomly assigned nephrologists within each site will receive the intervention (training to use the BC/WC tool) or to be in the waitlist control, meaning that they will not be offered BC/WC training until the end of the study, when all participants have been enrolled. Participants will be on follow up with surveys and chart review for up to two years after study enrollment. Caregivers will also be invited to participate and complete surveys.

DETAILED DESCRIPTION:
This study will test the effect of the Best Case/Worst Case intervention on receipt of palliative care and intensity of treatment at the end of life, quality of life, and quality of communication for older patients with end-stage renal disease (ESRD). This multi-site cluster randomized trial will enroll 320 participants who are making a dialysis initiation decision and receive care from a nephrologist trained to use the Best Case/Worst Case tool, or care from a nephrologist who has not been trained to use this tool (usual care). Randomly assigned nephrologists within each site will receive the intervention or waitlist control (upon study completion). Participants will be on follow up for up to two years after study enrollment via regular surveys and chart review. This study has three aims:

Aim 1: To test the effect of the Best Case/Worst Case intervention on (1) receipt of palliative care and (2) intensity of treatment at the end of life for older patients with ESRD. Chart reviews will be used to determine whether participants have received at least one outpatient or inpatient palliative care consultation within 12 months of enrollment in the study. These consultations must be clearly marked as palliative care, provided by a clinician with palliative care training and have documented discussion of goals clarification, advance care planning, symptom management, coping, spiritual needs, or end-of-life care. To measure intensity of treatment received at the end of life, it will be determined whether participants have had an ICU admission within 30 days of death as a primary outcome and ICU admission, emergency room (ER) visit, or hospital admission within 30 days of death as a composite secondary outcome.

Aim 2: To test the effect of the Best Case/Worst Case intervention on quality of life. The primary outcome for Aim 2 is quality of life as measured by the Functional Assessment of Chronic Illness Therapy -Palliative Care (FACIT-Pal Version 4) at baseline, and every three months for up to 2 years after study enrollment. The hypothesis is that the overall quality of life will decline over time as participants become more infirm. The average change in health-related quality of life over time which has been shown to decline less with the receipt of concurrent palliative care will be compared.

Aim 3: To test the effect of the Best Case/Worst Case intervention on the quality of communication. To evaluate participant's assessment of nephrologist communication, the Quality of Communication (QOC) scale developed by Randy Curtis will be used. Unlike other measurements of physician communication that have high ceiling effects and limited ability to measure change, the QOC includes 7 items specific to end-of-life communication, which, if not performed by the clinician, are scored as zero. This will allow us to discriminate between quality of communication attributable to participant satisfaction (with high ceiling effects) versus content.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (eGFR) of less than or equal to 24
* Not currently on dialysis (participants are eligible if they have had intermittent dialysis in the past or have dialysis access in place but are not currently on dialysis)
* Participants must meet one or more of the following criteria: age greater than 80, evidence from the medical record that the patient has comorbid illness such that the modified Charlson score is 4 or greater, or a negative response to the standard "Surprise Question" ("Would you be surprised if this patient died in the next year?") from the participant's nephrologist.

Exclusion Criteria:

* Currently on dialysis
* Lack decision-making capacity
* Do not speak English

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Receipt of palliative care consult within 12 months of study enrollment, as determined by chart review or report by patient or caregiver | from enrollment up to 12 months, data collected up to 2 years
  Number of patients with 1 or more palliative care consults within 12 months of study enrollment.

SECONDARY OUTCOMES:
Receipt of palliative care during 2-year follow up as determined by chart review or report by patient or caregiver | From enrollment for up to 2 years
  Number of patients with receipt of any palliative care as determined by chart review or patient or caregiver report during 2-year follow up.
Patient-reported health-related quality of life | Every 3 months for up to 2 years after enrollment
  Patient-reported health related quality of life will be measured using the 46-item Functional Assessment of Chronic Illness Therapy-Palliative Care Version 4 (FACIT-Pal); the investigators will compare the average score and average change (slope) in health-related quality of life over time, using the total score at last follow up. Possible scores for the FACIT-Pal total score range from 0-184. Higher scores indicate better quality of life.
Patient-reported health-related quality of life | Every 3 months for up to 2 years after enrollment
  Patient-reported health related quality of life will be measured using the 27-item Functional Assessment of Cancer Therapy - General (FACT-G) scale (used here in non-cancer patients as part of the FACIT-Pal instrument). Possible scores for the FACT-G total score range from 0-108. Higher scores indicate better quality of life.
Patient-reported health-related quality of life | Every 3 months for up to 2 years after enrollment
  Patient-reported health related quality of life will be measured using the 19-item FACIT-Pal palliative care subscale (PalS). Possible scores for the PalS range from 0-76. Higher scores indicate better quality of life.
Patient-reported quality of communication (QOC) received from study nephrologist | 48 hours after enrollment
  Patient-reported general quality of communication will be measured using the 19-item Quality of Communication (QOC) scale. The QOC is a validated self-report instrument. The average composite score will be given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication.
Patient-reported general quality of communication (QOC) received from study nephrologist | 48 hours after enrollment
  Patient-reported general quality of communication will be measured using the 6-item general communication subscale of the 19-item Quality of Communication (QOC) scale. The QOC is a validated self-report instrument. The average item score will be given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication.
Patient-reported quality of end-of-life communication (QOC) received from study nephrologist | 48 hours after enrollment
  Patient-reported quality of end-of-life communication will be measured using 7-item end-of-life communication subscale of the 19-item Quality of Communication scale. The QOC is a validated self-report instrument. The average item score will be given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication.
Hospice enrollment during 2-year follow up as determined by chart review or report by patient or caregiver | From enrollment for up to 2 years
  Number of patients with documentation of hospice enrollment as determined by chart review and patient or caregiver report during 2-year follow up.
Documentation of new advance care planning during 2-year follow up as determined by chart review or report by patient or caregiver | From enrollment for up to 2 years
  Number of patients with new documentation of advance care planning as determined by chart review or patient or caregiver report during 2-year follow up.
Treatment intensity at the end of life review as determined by chart review or report by patient or caregiver | Within 30 days of death
  Number of patients with one or more of the following within 30 days of death: ER visit, ICU stay or hospitalization as determined by chart review or patient or caregiver report.
Surgical treatment intensity at the end of life as determined by chart review or report by patient or caregiver | Within 30 days of death
  Number of patients who had one or more surgical procedure within 30 day as determined by chart review or patient or caregiver report.
Initiation of dialysis as determined by chart review or report by patient or caregiver | From enrollment for up to 2 years
  Number of patients initiating dialysis as determined by chart review or patient or caregiver report.
Time to on-study death | From enrollment for up to 2 years
  Time, in six month intervals, from baseline to 2 years. The Kaplan-Meier estimate reports the percentage of participants who experience death within 2 years from randomization. Participant death will be ascertained through medical record review and caregiver report.
Caregiver-reported quality of dying and death | 3 months after death
  Quality of dying and death as perceived by the patient's caregiver will be measured using the Quality of Death and Dying (QODD) survey that asks about the patient's final 30 days of life. Possible scores on this measure range from 0 to 100 and higher scores indicate higher quality of dying and death.
Caregiver-reported health related quality of life | Every 3 months for up to 2 years after enrollment
  Caregiver-reported health related quality of life will be measured using the Cambridge Palliative Audit Schedule (CAMPAS-R). Possible scores on this survey range from 0-100 and higher scores indicate greater symptomology.
Caregiver-reported general quality of communication (QOC) received from study nephrologist | Within 48 hours after enrollment
  Caregiver-reported general quality of communication will be measured using the 6-item general communication subscale of the 19-item Quality of Communication (QOC) scale. The QOC is a validated self-report instrument. Possible scores on this subscale range from 0-60. Higher scores indicate higher perceived quality of communication.
Caregiver-reported quality of end-of-life communication (QOC) received from study nephrologist | Within 48 hours after enrollment
  Caregiver-reported quality of end-of-life communication will be measured using 7-item end-of-life communication subscale of the 19-item Quality of Communication scale. The QOC is a validated self-report instrument. Possible scores on this subscale range from 0-70. Higher scores indicate higher perceived quality of communication.
Treatment intensity at the end of life as determined by chart review or report by patient or caregiver | Within 30 days before death
  Number of patients with 1 or more ICU admission within 30 days of death.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L Schwarze, MD, MPP, FACS, Principal Investigator — University of Wisconsin, Madison; Amar Bansal, MD, Principal Investigator — University of Pittsburgh; Katharine Cheung, MD, PhD, Principal Investigator — University of Vermont; Deidra Crews, MD, Principal Investigator — Johns Hopkins University; Katie Colborn, PhD, Principal Investigator — University of Colorado, Denver; Holly Koncicki, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jean Kutner, MD, Principal Investigator — University of Colorado, Denver; Daniel Lam, MD, Principal Investigator — University of Washington; Alvin Moss, MD, Principal Investigator — West Virginia University; Maya Rao, MD, Principal Investigator — Columbia University; Dawn Wolfgram, MD, Principal Investigator — Medical College of Wisconsin; Jeniann Yi, MD, Principal Investigator — University of Colorado, Denver; Tamara Isakova, MD, MMSc, Principal Investigator — Northwestern University
Locations (11):
- United States (11):
  - University of Colorado, Denver, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Department of Medicine, University of Vermont, Burlington, Vermont
  - University of Washington, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data set from this project will be stored in the Palliative Care Research Cooperative Group (PCRC) De-identified Data Repository (DiDR).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year after study completion or two months after initial manuscript has been accepted for publication (whichever comes first), UW will securely transfer a de-identified dataset to the PCRC Data Repository.
Access Criteria: Investigators may request access to de-identified study data for secondary analyses using the PCRC Data Repository webform. Requests must include a summary of the following: research questions, objectives, hypotheses, statistical analysis plan, and project timeline. Requestors must provide a list of specific variables they would like included in the secondary data set. Each request must also include a data security plan and explanation of how the data will be stored and who will have access to it. The PCRC staff and UW PI will review all requests assessing the scientific integrity, feasibility and analytic rigor.
URL: https://palliativecareresearch.org/corescenters/data-informatics-statistics-core-disc/pcrc-de-identified-data-repository-didr

REFERENCES:
- [Background] Schell JO, Patel UD, Steinhauser KE, Ammarell N, Tulsky JA. Discussions of the kidney disease trajectory by elderly patients and nephrologists: a qualitative study. Am J Kidney Dis. 2012 Apr;59(4):495-503. doi: 10.1053/j.ajkd.2011.11.023. Epub 2012 Jan 4. PMID 22221483
- [Background] Ladin K, Lin N, Hahn E, Zhang G, Koch-Weser S, Weiner DE. Engagement in decision-making and patient satisfaction: a qualitative study of older patients' perceptions of dialysis initiation and modality decisions. Nephrol Dial Transplant. 2017 Aug 1;32(8):1394-1401. doi: 10.1093/ndt/gfw307. PMID 27576590
- [Derived] Haug K, Buffington A, Zelenski A, Hanlon BM, Stalter L, Kwekkeboom KL, Rathouz P, Bansal AD, Cheung K, Crews D, Frazier R, Koncicki H, Lam D, Moss A, Rao M, Wolfgram DF, Yi J, Brill C, Kendrick R, Campbell TC, Jhagroo R, Schwarze M. Best Case/Worst Case: protocol for a multisite randomised clinical trial of a scenario planning intervention for patients with kidney failure. BMJ Open. 2022 Nov 3;12(11):e067258. doi: 10.1136/bmjopen-2022-067258. PMID 36328383

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT04466865/SAP_004.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04466865/ICF_005.pdf